CLINICAL TRIAL: NCT06780280
Title: Walking With Overground Robotic Exoskeletons to Improve Arrousal in Individuals With Disorders of Consciousness
Acronym: ORE-DOC
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Craig Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-2874
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Traumatic Brain Injuries
Keywords: TBI, disorders of consciousness, walking, exoskeletons
MeSH Terms: conditions — Brain Injuries, Traumatic; Consciousness Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Walking Intervention (Experimental): Overground walking with an exoskeleton
  Interventions: Other: Overground Walking

INTERVENTIONS:
Other: Overground Walking — Overground walking with an exoskeleton

SUMMARY:
This proposed study will examine a walking intervention to promote changes in conscious state in individuals with disorders of consciousness (DoC) due to acquired brain injury (ABI). Recent practice guidelines highlight the need to develop interventions to arouse patients with DoC, as current treatment options are scarce with limited to low-quality pharmaceutical and electrical stimulation approaches to improve outcomes. New data indicates patients with chronic DoC may benefit from therapeutic intervention prioritizing repeated multimodal sensory (i.e., simultaneous vestibular, proprioceptive, and visual) input, but likely not attain comparable functional recovery to those who demonstrate early command following ability. Interventions activating pathways of the cerebral consciousness network may leverage a substrate for recovery. We hypothesize that walking in an overground robotic exoskeleton (ORE) is safe, feasible, and will simultaneously stimulate endogenous cognitive and automatic pathways associated with walking5 to promote changes in behavioral performance in individuals with DoC.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the safety, feasibility and tolerability of using ORE therapy with individuals who meet criteria for DoC during inpatient rehabilitation while evaluating changes in behavioral performance, neurophysiology, and physiologic response to training. DoC numbers are very small so our goal is to gather this pilot data to support a future multi-site efficacy study with other TBIMS Center partners.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with DOC who are receiving inpatient rehabilitation

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events and feasibility | four weeks
  We will measure all adverse advents.

SECONDARY OUTCOMES:
Coma Recovery Scale-Revised | four weeks
  Measuring motor subscale, arrousal, and auditory subscales

IPD SHARING:
Plan to Share IPD: No
Pilot study